CLINICAL TRIAL: NCT06345547
Title: Prospective Observational Cohort Survey to Assess the Prevalence and Development of Sarcopenia and the Correlation of Muscle Mass and Outcome in Patients with Cirrhosis by Skeletal Muscle Ultrasound.
Brief Title: Muscle Mass Via UltraSound in Cirrhosis (MMUSCLE)
Acronym: MMUSCLE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Karolien Dams, Principal Investigator, MD, senior staff intensive care, University Hospital, Antwerp
Other Study IDs: EDGE 003539
Record Dates: First submitted 2024-03-14; First posted 2024-04-03 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Sarcopenia; Cirrhosis; Malnutrition
Keywords: sarcopenia; cirrhosis; malnutrition; skeletal muscle ultrasound
MeSH Terms: conditions — Sarcopenia; Fibrosis; Malnutrition | interventions — High-Energy Shock Waves; Hand Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Child A: The impact of sarcopenia in patients with cirrhosis may also be influenced by sex, severity of hepatic dysfunction, and etiology of cirrhosis. For this reason we aim for an homogeneous population, with a balanced distribution over the Child Pugh classification with a homogeneous population of at least 50%.
  Child A patients still have a good hepatic function.
  Interventions: Other: ultrasound
- Child B: Child B patients have a moderately impaired hepatic function.
  Interventions: Other: ultrasound
- Child C: Patients with Child C have an advanced hepatic dysfunction, within this group we will also look at patients with acute on chronic liver failure.(ACLF)
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — Ultrasound of m. quadriceps and m. thenar All ultrasound measurements will be performed in triplicate, with the average of the scores used in final analyses. Four parameters will be evaluated: muscle thickness, muscle cross sectional area, pennation angle and echo intensity (gain, depth and frequency will be kept constant).
  Hand grip strength measurement: measurement by an electronic hand dynamometer DynEx1TM (MD Systems, Inc. Ohio, USA). The recommendations for the handgrip strength test of the American Society of Hand Therapists will be followed: The maximum of the three values will be considered for analysis.
  Other Names: hand grip strength

SUMMARY:
The goal of this observational cohort study is to learn about loss of muscle mass and muscle strength (sarcopenia) in patients with cirrhosis. The main question[s] it aims to answer are:

* what is the prevalence and development of sarcopenia in cirrhosis?
* what is the role of malnutrition? Participants will

  * undergo a muscle ultrasound of the lower and upper limb muscles
  * handgrip strength will be measured
  * malnutrition screening and assessment
  * complete a questionnaire to assess quality of life

DETAILED DESCRIPTION:
In this study, the investigators will assess the prevalence and development of sarcopenia in the large in- and outpatient population with cirrhosis (n= 1346) of the University Hospital of Antwerp, using ultrasound assessment of muscle mass and quality in the lower as well as the upper limb muscles. Handgrip strength will be tested for muscle functional status. Findings will be correlated with clinical outcome (MELD, survival, decompensating events). The etiology of the cirrhosis and its underlying activity will be taken into account as dependent variables, e.g. whether there is a difference between compensated vs. decompensated cirrhosis. The investigators will screen for malnutrition using the RFH-NPT and compare with the GLIM criteria. The effect of sarcopenia on the quality of life will be evaluated using the validated "SarQoL®" (Sarcopenia Quality of Life) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cirrhosis and follow-up in the University Hospital of Antwerp

Exclusion Criteria:

* known patient will against participation in the study or against the measures applied in the study
* a decision made prior to inclusion to stop further treatment of the patient within the next 24 hours
* no complete remission of malignancy including hepatocellular carcinoma within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From our large population we will prospectively evaluate 60 patients with all 3 muscle parameters (US m quadriceps, US m thenar and hand grip strength). This will allow to calculate the incidence rate and relative risk of sarcopenia presence in this population. To keep the population homogeneous we will include patients according to the Child-Pugh classification with a balanced distribution between the subclasses.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sarcopenia: muscle mass | baseline
  Number of patients with prevalent sarcopenia. This will be assessed by skeletal muscle ultrasound (muscle thickness expressed in cm).
  Sarcopenia has been defined by the European Working Group on Sarcopenia as "a progressive and generalized skeletal muscle disorder associated with an increased likelihood of adverse outcomes including falls, fractures, disability, and mortality," combining both muscle mass and muscle strength or muscle performance in its definition. This first outcome measure defines muscle mass.
Prevalence of sarcopenia: muscle strength | baseline
  Number of patients with prevalent sarcopenia. This will be assessed by handgrip strength (expressed in kg).
  Sarcopenia has been defined by the European Working Group on Sarcopenia as "a progressive and generalized skeletal muscle disorder associated with an increased likelihood of adverse outcomes including falls, fractures, disability, and mortality," combining both muscle mass and muscle strength or muscle performance in its definition.
  As the definition contains both muscle mass and muscle strength, both factors have to be evaluated. This second outcome measure defines muscle strength.
Development of sarcopenia: changes in muscle mass | 2 years
  Changes in muscle mass by ultrasound muscle parameters from baseline up to 2 years follow-up. We will evaluate the muscle parameters that define muscle mass: muscle thickness expressed in cm, cross sectional area in squared cm, pennation angle in degrees and echo intensity expressed in arbitrary units (A.U.)
Development of sarcopenia: changes in muscle strength | 2 years
  This will be assessed by handgrip strength (expressed in kg). Sarcopenia has been defined by the European Working Group on Sarcopenia as "a progressive and generalized skeletal muscle disorder associated with an increased likelihood of adverse outcomes including falls, fractures, disability, and mortality," combining both muscle mass and muscle strength or muscle performance in its definition.
  As the definition contains both muscle mass and muscle strength, both factors have to be evaluated.
Development of sarcopenia: changes in muscle quality | 2 years
  Changes in muscle mass by ultrasound muscle parameters from baseline up to 2 years follow-up. We will evaluate the muscle parameters that define quality of muscle: pennation angle in degrees and echo intensity expressed in arbitrary units (A.U.)

SECONDARY OUTCOMES:
Decompensation events: MELD score • MELD evolution | 2 years
  clinical evolution of cirrhosis: MELD (Model of Endstage Liver Disease) score in points (range 7-40), with a higher score defining a worse state.
Decompensation events: mortality • MELD evolution | 2 years
  clinical evolution of cirrhosis: Mortality 1 year after enrolment (Y/N)
Decompensation events: transplantation • MELD evolution | 2 years
  clinical evolution of cirrhosis: Need for transplantation/transplant outcome (Y/N)
Malnutrition | 2 years
  The European Society for Clinical Nutrition and Metabolism guidelines recommend the Royal Free Hospital-Nutritional Prioritizing Tool (RFH-NPT) to identify malnutrition risk in patients with liver disease. The RFH-NPT categorises nutritional risk as low (0 points), medium (1 points) and high (2-7 points).
  The Global Leadership Initiative on Malnutrition (GLIM) has established a global consensus on the criteria for diagnosing malnutrition in adults in hospital settings. It is a two-step approach for the malnutrition diagnosis, i.e., first screening to identify "at risk" status by the use of any validated screening tool, and second, assessment for diagnosis and grading the severity of malnutrition; mild - moderate - severe.
Quality of life in cirrhosis | 2 years
  The effect of sarcopenia on the quality of life will be evaluated using the validated SarQoL® questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Karolien Dams, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data that underlie the results reported in the article, after deidentification (text, table, figures, appendices).

REFERENCES:
- [Background] Dhaliwal A, Armstrong MJ. Sarcopenia in cirrhosis: A practical overview. Clin Med (Lond). 2020 Sep;20(5):489-492. doi: 10.7861/clinmed.2020-0089. PMID 32934043
- [Background] Lai JC, Tandon P, Bernal W, Tapper EB, Ekong U, Dasarathy S, Carey EJ. Malnutrition, Frailty, and Sarcopenia in Patients With Cirrhosis: 2021 Practice Guidance by the American Association for the Study of Liver Diseases. Hepatology. 2021 Sep;74(3):1611-1644. doi: 10.1002/hep.32049. No abstract available. PMID 34233031
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Hsu CS, Kao JH. Sarcopenia and chronic liver diseases. Expert Rev Gastroenterol Hepatol. 2018 Dec;12(12):1229-1244. doi: 10.1080/17474124.2018.1534586. Epub 2018 Oct 16. PMID 30791794
- [Background] Carey EJ, Lai JC, Sonnenday C, Tapper EB, Tandon P, Duarte-Rojo A, Dunn MA, Tsien C, Kallwitz ER, Ng V, Dasarathy S, Kappus M, Bashir MR, Montano-Loza AJ. A North American Expert Opinion Statement on Sarcopenia in Liver Transplantation. Hepatology. 2019 Nov;70(5):1816-1829. doi: 10.1002/hep.30828. Epub 2019 Aug 19. PMID 31220351
- [Background] Tandon P, Low G, Mourtzakis M, Zenith L, Myers RP, Abraldes JG, Shaheen AA, Qamar H, Mansoor N, Carbonneau M, Ismond K, Mann S, Alaboudy A, Ma M. A Model to Identify Sarcopenia in Patients With Cirrhosis. Clin Gastroenterol Hepatol. 2016 Oct;14(10):1473-1480.e3. doi: 10.1016/j.cgh.2016.04.040. Epub 2016 May 14. PMID 27189915
- [Background] Watanabe Y, Yamada Y, Fukumoto Y, Ishihara T, Yokoyama K, Yoshida T, Miyake M, Yamagata E, Kimura M. Echo intensity obtained from ultrasonography images reflecting muscle strength in elderly men. Clin Interv Aging. 2013;8:993-8. doi: 10.2147/CIA.S47263. Epub 2013 Jul 25. PMID 23926426
- [Background] Perkisas S, Baudry S, Bauer J, Beckwee D, De Cock AM, Hobbelen H, Jager-Wittenaar H, Kasiukiewicz A, Landi F, Marco E, Merello A, Piotrowicz K, Sanchez E, Sanchez-Rodriguez D, Scafoglieri A, Cruz-Jentoft A, Vandewoude M. Application of ultrasound for muscle assessment in sarcopenia: towards standardized measurements. Eur Geriatr Med. 2018 Dec;9(6):739-757. doi: 10.1007/s41999-018-0104-9. Epub 2018 Sep 17. PMID 34674473
- [Background] Stock MS, Thompson BJ. Echo intensity as an indicator of skeletal muscle quality: applications, methodology, and future directions. Eur J Appl Physiol. 2021 Feb;121(2):369-380. doi: 10.1007/s00421-020-04556-6. Epub 2020 Nov 21. PMID 33221942
- [Background] Iacob S, Mina V, Mandea M, Iacob R, Vadan R, Boar V, Ionescu G, Buzescu D, Gheorghe C, Gheorghe L. Assessment of Sarcopenia Related Quality of Life Using SarQoL(R) Questionnaire in Patients With Liver Cirrhosis. Front Nutr. 2022 Feb 25;9:774044. doi: 10.3389/fnut.2022.774044. eCollection 2022. PMID 35284449
- [Background] Perkisas S, Bastijns S, Baudry S, Bauer J, Beaudart C, Beckwee D, Cruz-Jentoft A, Gasowski J, Hobbelen H, Jager-Wittenaar H, Kasiukiewicz A, Landi F, Malek M, Marco E, Martone AM, de Miguel AM, Piotrowicz K, Sanchez E, Sanchez-Rodriguez D, Scafoglieri A, Vandewoude M, Verhoeven V, Wojszel ZB, De Cock AM. Application of ultrasound for muscle assessment in sarcopenia: 2020 SARCUS update. Eur Geriatr Med. 2021 Feb;12(1):45-59. doi: 10.1007/s41999-020-00433-9. Epub 2021 Jan 2. PMID 33387359
- [Background] Misirlioglu TO, Ozyemisci Taskiran O. Reliability of sonographic muscle thickness measurements of the thenar and hypothenar muscles. Muscle Nerve. 2018 Jan;57(1):E14-E17. doi: 10.1002/mus.25735. Epub 2017 Jul 18. PMID 28662294
- [Background] Pedrianes-Martin PB, Hernanz-Rodriguez GM, Gonzalez-Martin JM, Perez-Valera M, De Pablos-Velasco PL. Ultrasonographic Size of the Thenar Muscles of the Nondominant Hand Correlates with Total Body Lean Mass in Healthy Subjects. Acad Radiol. 2021 Apr;28(4):517-523. doi: 10.1016/j.acra.2020.02.029. Epub 2020 Jul 30. PMID 32739076
- [Background] Lopes J, Grams ST, da Silva EF, de Medeiros LA, de Brito CMM, Yamaguti WP. Reference equations for handgrip strength: Normative values in young adult and middle-aged subjects. Clin Nutr. 2018 Jun;37(3):914-918. doi: 10.1016/j.clnu.2017.03.018. Epub 2017 Mar 24. PMID 28389120